CLINICAL TRIAL: NCT03148145
Title: Mobile Phone-Based Physical Activity Intervention on University Staff
Brief Title: CalFitness Smartphone-Delivered Physical Activity Intervention With Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Anil Aswani, Assistant Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-03-8609
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Sedentary Lifestyle; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Constant Steps Goal (Active Comparator): Step Goal Delivery by Smartphone
  Interventions: Behavioral: Step Goal Delivery by Smartphone
- Averaged Steps Goals and Random Messages (Experimental): Step Goal Delivery by Smartphone Message Delivery by Smartphone
  Interventions: Behavioral: Step Goal Delivery by Smartphone; Behavioral: Message Delivery by Smartphone
- Algorithm Steps Goal and Random Messages (Experimental): Step Goal Delivery by Smartphone Message Delivery by Smartphone
  Interventions: Behavioral: Step Goal Delivery by Smartphone; Behavioral: Message Delivery by Smartphone
- Algorithm Steps Goal and Messages (Experimental): Step Goal Delivery by Smartphone Message Delivery by Smartphone
  Interventions: Behavioral: Step Goal Delivery by Smartphone; Behavioral: Message Delivery by Smartphone

INTERVENTIONS:
Behavioral: Step Goal Delivery by Smartphone — Step Goal Delivery by Smartphone
Behavioral: Message Delivery by Smartphone — Message Delivery by Smartphone
  Arms: Algorithm Steps Goal and Messages; Algorithm Steps Goal and Random Messages; Averaged Steps Goals and Random Messages

SUMMARY:
The overall goal of this study is to test personalized mobile phone-based physical activity interventions among students at the University of California, Berkeley. Most physical fitness applications for smartphones and activity trackers use a constant goal for the number of steps each day. However, if the step goals are dynamically adjusted according to past behavior, then the corresponding goals may encourage individuals to increase their physical activity level. This study consists of a randomized controlled trial in which we are assessing the efficacy of four different algorithms for calculating personalized goals for the number of steps each day and for determining which motivational messages to send each day.

ELIGIBILITY:
Inclusion Criteria:

* intent to become physically active
* own an iPhone 5s (or newer model)
* willing to keep the iPhone in pockets during the day
* willing to install and use the intervention app every day for 4 months
* ability to speak and read English.

Exclusion Criteria:

* known medical conditions or physical problems that require special attention in an exercise program
* planning an international trip during the next 4 months, which could interfere with daily server uploads of mobile phone data
* pregnant/gave birth during the past 6 months
* severe hearing or speech problem
* history of an eating disorder
* current substance abuse
* current participation in lifestyle modification programs or research studies that may confound study results
* history of bariatric surgery or plans for bariatric surgery in the next 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Daily Steps Taken Per Day | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States